CLINICAL TRIAL: NCT00715273
Title: Carotid Plaque Composition by Magnetic Resonance Imaging During Lipid Lowering Therapy
Brief Title: Evaluate Carotid Artery Plaque Composition by Magnetic Resonance Imaging in People Receiving Cholesterol Medication
Acronym: CPC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Pfizer (Industry); Abbott (Industry); Daiichi Sankyo (Industry); Upsher-Smith Laboratories (Industry)
Responsible Party: Principal Investigator, Xue-Qiao Zhao, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: STUDY00001165; R01HL063895-05A1 (NIH)
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Results first posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-05

CONDITIONS: Coronary Artery Disease; Carotid Artery Diseases; Atherosclerosis
Keywords: Magnetic Resonance Imaging; Atherosclerotic Plaque; Lipid Lowering Therapy
MeSH Terms: conditions — Coronary Artery Disease; Carotid Artery Diseases; Atherosclerosis; Plaque, Atherosclerotic | interventions — Atorvastatin; Niacin; Colesevelam Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- 1 - single therapy group (Active Comparator): Participants will receive atorvastatin, placebo niacin, and placebo colesevelam. The treatment target for LDL-C will be ≤80 mg/dl for the single therapy group.
  Interventions: Drug: Atorvastatin; Drug: Placebo Niacin; Drug: Placebo Colesevelam
- 2 - double therapy group (Experimental): Participants will receive atorvastatin, niacin, and placebo colesevelam. The treatment target for LDL-C will be ≤80 mg/dl for the double therapy group.
  Interventions: Drug: Atorvastatin; Drug: Niacin; Drug: Placebo Colesevelam
- 3 - triple therapy group (Experimental): Participants will receive atorvastatin, niacin, and colesevelam. The treatment target for LDL-C will be ≤60 mg/dl for the triple therapy group
  Interventions: Drug: Atorvastatin; Drug: Niacin; Drug: Colesevelam

INTERVENTIONS:
Drug: Atorvastatin — 10 to 80 mg of atorvastatin each day
  Other Names: Lipitor
Drug: Niacin — 2000 mg of niacin each day
  Other Names: Niaspan; Slo-niacin
  Arms: 2 - double therapy group; 3 - triple therapy group
Drug: Colesevelam — 3.8 g of colesevelam each day
  Other Names: WelChol
  Arms: 3 - triple therapy group
Drug: Placebo Niacin — Placebo niacin each day
  Arms: 1 - single therapy group
Drug: Placebo Colesevelam — Placebo colesevelam each day
  Arms: 1 - single therapy group; 2 - double therapy group

SUMMARY:
Atherosclerosis is a condition that occurs when fatty deposits build up along the inner walls of arteries. This study will examine the effectiveness of a combination of cholesterol-lowering medications at decreasing the fat content of atherosclerotic deposits in people who have coronary artery disease or carotid artery disease.

DETAILED DESCRIPTION:
Atherosclerosis is a condition in which deposits of fat, cholesterol, and other substances build up along the inner walls of arteries; these deposits are known as plaque. People with atherosclerosis are at risk of developing coronary artery disease, in which plaque build-up occurs in the arteries that supply blood to the heart, and carotid artery disease, in which plaque build-up occurs in the arteries that deliver blood through the neck to the brain. These conditions can lead to blood clots, heart attack, and stroke. Research has shown that people who have more fat content in atherosclerotic plaque may have a higher risk of experiencing a heart attack or stroke. Treatments for atherosclerosis include lifestyle changes, medicines, and medical procedures or surgery. There are several medications that can aid people in controlling their cholesterol levels, including atorvastatin, a medication that inhibits the production of cholesterol; niacin, a B-complex vitamin that can reduce cholesterol levels in combination with dietary changes; and colesevelam, a medication that inhibits fat absorption. Using magnetic resonance imaging (MRI), this study will evaluate whether these medications, alone or in combination, can decrease the fat content of atherosclerotic plaques within the carotid arteries of people with coronary artery disease and carotid artery disease.

This study will enroll people with coronary artery disease or carotid artery disease. Participants will be randomly assigned to one of the following 40-month treatment groups:

* Group 1 participants will receive atorvastatin, placebo niacin, and placebo colesevelam each day.
* Group 2 participants will receive atorvastatin, niacin, and placebo colesevelam each day.
* Group 3 participants will receive atorvastatin, niacin, and colesevelam each day.

At a baseline study visit, participants will undergo a blood collection and will receive dietary counseling that will focus on lowering cholesterol levels. They will also undergo an MRI scan of their carotid arteries. For the next 4 months, participants will attend monthly study visits for repeat blood collection and dietary counseling; for the subsequent 36 months, participants will attend study visits every other month. Repeat carotid artery MRI scans will occur at Months 12, 24, and 36. At three different times during the study, researchers will ask participants to record their food consumption for 3 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Clinically established coronary artery disease or carotid artery disease with greater than 15% stenosis by ultrasound
* Family history of cardiovascular disease
* Apolipoprotein B level greater than or equal to 120 mg/dL (LDL level should be between 100 and 190 mg/dL without medication)
* Has been undergoing lipid therapy for no more than 12 months before study entry
* Medically stable
* Medically able to undergo MRI procedure

Exclusion Criteria:

* Uses pacemaker or has metallic implants
* Has immediate plans for carotid endarterectomy
* History of alcohol or drug abuse
* Active liver disease or liver dysfunction, defined by elevations in alanine aminotransferase (ALT)/aspartate aminotransferase (AST) levels greater than 1.5 times the upper limit of normal
* Serum creatine kinase (CK) level greater than 3 times the upper limit of normal before study entry
* Serum creatinine level greater than 2.5 times the upper limit of normal
* Diabetes, with a fasting glucose level greater than 150 mg/dL or hemoglobin A1c (HbA1c) level greater than 8% before study entry
* Uncontrolled high blood pressure, defined as average resting systolic blood pressure greater than 200 mm Hg or average resting diastolic blood pressure greater than 95 mm Hg

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2001-05-01 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2019-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xue-Qiao Zhao, MD, Principal Investigator — University of Washington
Locations (4):
- United States (4):
  - University of Southern California, Los Angeles, California
  - St. Luke's Idaho Cardiology, Boise, Idaho
  - University of Washington Coronary Atherosclerosis Research Lab, Seattle, Washington
  - Yakima Heart Center, Yakima, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhao XQ, Phan BA, Chu B, Bray F, Moore AB, Polissar NL, Dodge JT Jr, Lee CD, Hatsukami TS, Yuan C. Testing the hypothesis of atherosclerotic plaque lipid depletion during lipid therapy by magnetic resonance imaging: study design of Carotid Plaque Composition Study. Am Heart J. 2007 Aug;154(2):239-46. doi: 10.1016/j.ahj.2007.04.035. PMID 17643572
- [Result] Moore A, Phan BA, Challender C, Williamson J, Marcovina S, Zhao XQ. Effects of adding extended-release niacin and colesevelam to statin therapy on lipid levels in subjects with atherosclerotic disease. J Clin Lipidol. 2007 Dec;1(6):620-5. doi: 10.1016/j.jacl.2007.09.001. Epub 2007 Sep 15. PMID 21291704
- [Result] Green PS, Vaisar T, Pennathur S, Kulstad JJ, Moore AB, Marcovina S, Brunzell J, Knopp RH, Zhao XQ, Heinecke JW. Combined statin and niacin therapy remodels the high-density lipoprotein proteome. Circulation. 2008 Sep 16;118(12):1259-67. doi: 10.1161/CIRCULATIONAHA.108.770669. Epub 2008 Sep 2. PMID 18765395
- [Result] Phan BA, Munoz L, Shadzi P, Isquith D, Triller M, Brown BG, Zhao XQ. Effects of niacin on glucose levels, coronary stenosis progression, and clinical events in subjects with normal baseline glucose levels (<100 mg/dl): a combined analysis of the Familial Atherosclerosis Treatment Study (FATS), HDL-Atherosclerosis Treatment Study (HATS), Armed Forces Regression Study (AFREGS), and Carotid Plaque Composition by MRI during lipid-lowering (CPC) study. Am J Cardiol. 2013 Feb 1;111(3):352-5. doi: 10.1016/j.amjcard.2012.09.034. Epub 2012 Nov 17. PMID 23168285
- [Result] Ronsein GE, Hutchins PM, Isquith D, Vaisar T, Zhao XQ, Heinecke JW. Niacin Therapy Increases High-Density Lipoprotein Particles and Total Cholesterol Efflux Capacity But Not ABCA1-Specific Cholesterol Efflux in Statin-Treated Subjects. Arterioscler Thromb Vasc Biol. 2016 Feb;36(2):404-11. doi: 10.1161/ATVBAHA.115.306268. Epub 2015 Dec 17. PMID 26681752
- [Result] Zhao XQ, Yuan C, Shah PK. Imaging to Assess the Effect of Anti-Inflammatory Therapy in Aortic and Carotid Atherosclerosis. J Am Coll Cardiol. 2016 Oct 18;68(16):1781-1784. doi: 10.1016/j.jacc.2016.08.011. No abstract available. PMID 27737745
- [Result] Chu MP, Many G, Isquith DA, McKeeth S, Williamson J, Neradilek MB, Colletti P, Zhao XQ. Metabolic and inflammatory risk reduction in response to lipid-lowering and lifestyle modification in the medically underserved individuals. Am J Prev Cardiol. 2021 Jul 31;7:100227. doi: 10.1016/j.ajpc.2021.100227. eCollection 2021 Sep. PMID 34401861
- [Result] Han T, Paramsothy P, Hong J, Isquith D, Xu D, Bai H, Neradilek M, Gill E, Zhao XQ. High-resolution MRI assessed carotid atherosclerotic plaque characteristics comparing men and women with elevated ApoB levels. Int J Cardiovasc Imaging. 2020 Mar;36(3):481-489. doi: 10.1007/s10554-019-01600-1. Epub 2020 Feb 4. PMID 32020410
- [Result] Zhao XQ, Dong L, Hatsukami T, Phan BA, Chu B, Moore A, Lane T, Neradilek MB, Polissar N, Monick D, Lee C, Underhill H, Yuan C. MR imaging of carotid plaque composition during lipid-lowering therapy a prospective assessment of effect and time course. JACC Cardiovasc Imaging. 2011 Sep;4(9):977-86. doi: 10.1016/j.jcmg.2011.06.013. PMID 21920335
- [Result] Dong L, Kerwin WS, Chen H, Chu B, Underhill HR, Neradilek MB, Hatsukami TS, Yuan C, Zhao XQ. Carotid artery atherosclerosis: effect of intensive lipid therapy on the vasa vasorum--evaluation by using dynamic contrast-enhanced MR imaging. Radiology. 2011 Jul;260(1):224-31. doi: 10.1148/radiol.11101264. Epub 2011 Apr 14. PMID 21493792
- [Result] Kerwin WS, Zhao X, Yuan C, Hatsukami TS, Maravilla KR, Underhill HR, Zhao X. Contrast-enhanced MRI of carotid atherosclerosis: dependence on contrast agent. J Magn Reson Imaging. 2009 Jul;30(1):35-40. doi: 10.1002/jmri.21826. PMID 19557844
- [Derived] Ronsein GE, Vaisar T, Davidson WS, Bornfeldt KE, Probstfield JL, O'Brien KD, Zhao XQ, Heinecke JW. Niacin Increases Atherogenic Proteins in High-Density Lipoprotein of Statin-Treated Subjects. Arterioscler Thromb Vasc Biol. 2021 Aug;41(8):2330-2341. doi: 10.1161/ATVBAHA.121.316278. Epub 2021 Jun 17. PMID 34134520

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1 - Single Therapy Group | 2 - Double Therapy Group | 3 - Triple Therapy Group
Started | 71 | 73 | 73
Completed | 63 | 65 | 68
Not Completed | 8 | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 - Single Therapy Group | 2 - Double Therapy Group | 3 - Triple Therapy Group | Total
Number analyzed (Participants) | 71 | 73 | 73 | 217
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 60 | 62 | 60 | 182
  >=65 years | 11 | 11 | 13 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 30 | 30 | 88
  Male | 43 | 43 | 43 | 129
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 12 | 10 | 31
  Not Hispanic or Latino | 62 | 61 | 63 | 186
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 3 | 3 | 5 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 2 | 5
  White | 65 | 65 | 64 | 194
  More than one race | 3 | 1 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 71 | 73 | 73 | 217
Family history of premature cardiovascular disease, n (%) [Count of Participants; unit: Participants] | 34 | 36 | 36 | 106
History of myocardial infarction, n (%) [Count of Participants; unit: Participants] | 25 | 26 | 31 | 82
Established coronary artery disease, n (%) [Count of Participants; unit: Participants] | 62 | 60 | 67 | 189
Hypertension, n (%) [Count of Participants; unit: Participants] | 42 | 44 | 44 | 130
Diabetes, n (%) [Count of Participants; unit: Participants] | 10 | 13 | 9 | 32
Current smoking, n (%) [Count of Participants; unit: Participants] | 13 | 17 | 15 | 45

OUTCOME MEASURES:

1. Primary Outcome: Annualized LRNC Volume Change in Carotid Plaque Composition, as Assessed by MRI
Description: The primary endpoint of this study is carotid plaque lipid composition identified by MRI. The determination of plaque lipid content for each carotid artery will be performed using the automated interactive system. These measurements will be performed from the MRI scans at four time points blinded to time sequence of MRI examinations, patient treatment, lipid levels and clinical course.
  Volume Measurements: Contours were placed around the lumen, outer-wall boundaries, and plaque features of carotid artery. (Arterial wall area) = (outer-wall area) - (lumen area). Volume calculated as: area x 2 mm (slice thickness). Tissue volume/wall volume x (100%) is presented as percentage. Annualized change presented mm^3/year (for volume) and as percentage change/year.
Time Frame: Measured at Years 1, 2, and 3
Population: Analysis group was limited from total study population due to the need for detectable lipid-rich necrotic core (LRNC) measurement at study baseline.
Measure: Mean (Standard Error); unit: mm^3/year
Arm/Group | 1 - Single Therapy Group | 2 - Double Therapy Group | 3 - Triple Therapy Group
Number analyzed (Participants) | 60 | 61 | 61
mm^3/year | -4.6 (5.0) | -15.1 (3.2) | -9.4 (3.0)

2. Secondary Outcome: Composite of Cardiovascular Endpoints: Number of Participants With Cardiovascular Disease Death, Non-fatal Heart Attack, Stroke, and Worsening Ischemia Requiring Medical Interventions
Description: Any cardiovascular events such as death from any cause, nonfatal myocardial infarction, stroke, and revascularization procedures (PCI or CABG) due to unstable ischemia will be recorded and verified.
Time Frame: Measured at Years 3, 4, and 5
Measure: Count of Participants; unit: Participants
Arm/Group | 1 - Single Therapy Group | 2 - Double Therapy Group | 3 - Triple Therapy Group
Number analyzed (Participants) | 71 | 73 | 73
Participants
  Composite Measured at Year 3 | 6 | 6 | 7
  Composite Measured at Year 4 (cumulative) | 7 | 11 | 9
  Composite Measured at Year 5 (cumulative) | 9 | 11 | 9

3. Primary Outcome: Annualized LRNC and Wall Volume Changes in Carotid Plaque Composition, as Assessed by MRI
Description: as for outcome 1
Time Frame: Measured at Years 1, 2, and 3
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage change/year
Arm/Group | 1 - Single Therapy Group | 2 - Double Therapy Group | 3 - Triple Therapy Group
Number analyzed (Participants) | 60 | 61 | 61
percentage change/year
  LRNC change | -1.6 (1.1) | -3.6 (0.8) | -2.8 (0.7)
  Wall Volume change | -0.6 (0.5) | -1.4 (0.4) | -1.2 (0.5)

ADVERSE EVENTS:
Time Frame: Period of time from study baseline visit until subject completion. Subject followed for up to 168 months in open label follow-up period.
Arm/Group | 1 - Single Therapy Group | 2 - Double Therapy Group | 3 - Triple Therapy Group
All-Cause Mortality (participants affected / at risk) | 7/71 | 7/73 | 3/73
Serious Adverse Events (participants affected / at risk) | 26/71 | 20/73 | 20/73
Other Adverse Events (participants affected / at risk) | 34/71 | 40/73 | 32/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 - Single Therapy Group (N=71) | 2 - Double Therapy Group (N=73) | 3 - Triple Therapy Group (N=73)
Myocardial infarction (Cardiac disorders) | 3 (3) | 4 (4) | 4 (4)
Stroke (General disorders) | 2 (2) | 1 (1) | 0 (0)
Coronary artery bypass graft surgery (Surgical and medical procedures) | 1 (1) | 2 (2) | 1 (1)
Percutaneous coronary intervention (Cardiac disorders) | 10 (13) | 6 (10) | 8 (8) — Single or multiple vessel
Peripheral artery revascularization (Vascular disorders) | 2 (3) | 2 (2) | 3 (3)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3) | 4 (4)
Hospitalized for worsening ischemia (Cardiac disorders) | 7 (9) | 7 (9) | 5 (6) — Hospitalization for worsening cardiac ischemia but no revascularization
Hospitalized for transient ischemic attack (Vascular disorders) | 2 (2) | 2 (2) | 1 (1)
Hospitalized for heart failure (Cardiac disorders) | 1 (2) | 0 | 1 (1)
Death - Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 2 (2)
Death - myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Death - Coronary artery disease (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Death - Intentional self-harm (General disorders) | 0 (0) | 0 (0) | 1 (1)
Death - Idiopathic Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Death - Other/Multiple/Unknown (General disorders) | 3 (3) | 2 (2) | 0 (0)
Diseased or injured hip joint requiring replacement (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 1 - Single Therapy Group (N=71) | 2 - Double Therapy Group (N=73) | 3 - Triple Therapy Group (N=73)
New onset Type 2 Diabetes Melitus (Endocrine disorders) | 4/61 (4) | 5/60 (5) | 3/64 (3)
Sinus infection (Infections and infestations) | 6 (6) | 0 (0) | 2 (2) — Sinus infection with or without antibiotic use
Muscle aches (General disorders) | 5 (5) | 1 (2) | 3 (3)
Leg pain (General disorders) | 2 (3) | 7 (7) | 6 (6)
Diseased or injured knee joint requiring surgery (Surgical and medical procedures) | 6 (6) | 3 (3) | 3 (3)
Headache (General disorders) | 5 (5) | 6 (6) | 2 (2)
Dizziness (General disorders) | 1 (1) | 9 (12) | 2 (2)
Kidney stone (Renal and urinary disorders) | 2 (2) | 0 (0) | 4 (5)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 4 (4) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 2 (2) | 5 (5) | 4 (4)
Upper respiratory infection (Infections and infestations) | 9 (13) | 11 (11) | 8 (10)
Influenza (Infections and infestations) | 3 (4) | 8 (10) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 7 (7)
Angina (Cardiac disorders) | 3 (4) | 9 (12) | 6 (8)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT00715273/Prot_SAP_000.pdf